CLINICAL TRIAL: NCT01867190
Title: An Open-label Single Arm Phase 2 Proof of Concept Study to Assess the Efficacy and Safety of ASCT01 in Patients With Critical Limb Ischemia
Brief Title: Study to Assess Efficacy and Safety of Bone Marrow Derived Stem Cells in Patients With Critical Limb Ischemia
Acronym: CLI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lifecells, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 15069
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Critical Limb Ischemia
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Autologous treatment for CLI open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ASCT01 (Other): ASCT01 (Autologous Stem Cell Transplantation)
  Interventions: Biological: ASCT01 (Autologous Stem Cell Transplantation)

INTERVENTIONS:
Biological: ASCT01 (Autologous Stem Cell Transplantation) — Single Administration of the entire ASCT01 preparation at rate if 10million CD45+ cells per milliliter at 5 ml per minute via the intra- via intra-arterial infusion route and 6 or more injections of approximately 0.2 ml each intramuscular route

SUMMARY:
This study will assess the safety and efficacy of intra-arterial infusion and intramuscular injection of an autologous, bone marrow-derived stem cell preparation (ASCT01) in patients with critical limb ischemia who have exhausted all medical and surgical therapeutic options. The safety and tolerability will be evaluated by regular monitoring of the general physical condition, vital signs, and the occurrence of AE and SAE, respectively. Furthermore, the standard biochemical and blood variables (red and white blood cell counts, Hb, Ht, platelets, sodium, potassium, chloride, calcium, phosphor, ASAT, ALAT, bilirubin, total protein, albumin, AP, cholesterol (LDL,HDL), triglycerides, urea and creatinine, immunoglobulins, HBA1c, C-peptide) will be checked before the treatment as well as 30 and 90 days after the treatment.

DETAILED DESCRIPTION:
Efficacy will be determined by number of collateral arteries as assessed magnetic resonance angiography at baseline and again at 3 months, rate of major amputation (above the ankle) of the affected limb within 3 months or an unchanged critical limb ischemia of the affected limb after 3 months defined as less than 15% change in tcPO2 or ABI or absolute ankle pressure.Efficacy endpoint is at 3 months. Clinical endpoints and safety will be measured through 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients in the age group of 18-80yrs.
2. Established CLI (confirmed by Rutherford 4 to 5) with angiographic evidence of significant infra-inguinal arterial occlusive disease
3. Ankle Brachial Pressure Index (ABI) ≤ 0.6 or the absolute ankle blood pressure < 60 mm Hg or TcPO2<20 mmHg without tissue loss or TcPO2<40 mmHg if there is tissue loss or alternatively toe Brachial Pressure Index (TBI) less 0.5 or the absolute toe blood pressure less than 50 mm Hg
4. No surgical or interventional option for revascularization and no response to best standard care delivered as confirmed by a vascular surgeon and/or physician.
5. No immediate life-threatening complication from CLI which would demand immediate amputation.
6. Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent, abide by the study requirements, and agree to return for required follow-up visits.
7. On optimal medical therapy
8. If diabetic, HgbA1c <10%

Exclusion Criteria:

1. Acute life threatening complication of limb ischemia with the need for immediate limb amputation to avoid death or clinical deterioration
2. Patients with confirmed Rutherford 6 condition with extensive tissue damage
3. Patients with documented terminal illness or cancer or any concomitant disease process with a life expectancy of less than 6 months.
4. Patients with a history of severe alcohol or drug abuse within 3 months of screening.
5. Known bone marrow diseases which preclude transplantation.
6. End-stage renal failure on regular dialysis treatment. Creatinine ≥2.0 mg/dl
7. Patients already enrolled in another investigational drug trial or completed within 1month.
8. Pregnancy.
9. Patients tested positive for HIV screen1or2, Hepatitis C antibody Hepatitis B surface-antigen, HepatitisBcore Antibody, Syphilis screen
10. Myocardial infarction / CVA / TIA within the past three months prior to enrollment
11. Revascularization procedure in target limb within 6 weeks prior to enrollment
12. Laboratory values as show below*
13. Currently taking immunosuppressive agents
14. If diabetic, diagnosis of proliferative retinopathy
15. Patients with infected ulcers or systemic infections *Laboratory Values: Hemoglobin <10 g/dL Platelet count <100,000/microL ALT >60 U/L AST >60 U/L Bilirubin >1.0 mg/dL INR >1.3 unless on Coumadin and at Investigator discretion APTT >40 second unless on Lovenox or Heparin and at Investigator's discretion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of intra-arterial infusion and intramuscular injection of ASCT01 on the combined primary endpoint of major amputation (above the ankle) or persisting critical limb ischemia (no clinical or perfusion improvement). | primary outcome measured at 3 months
  The primary outcome variable is "treatment failure" defined as major amputation (above the ankle) of the affected limb within 3 months or an unchanged critical limb ischemia of the affected limb after 3 months defined as less than 15% change in tcPO2 or ABI or absolute ankle pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Sudhakar, MS, Pharm, Study Director — Lifecells, LLC.
Locations (1):
- Kansas City Vascular Foundation (KCV), North Kansas City, Missouri, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT01867190/Prot_SAP_000.pdf